CLINICAL TRIAL: NCT02983695
Title: Cannabinoid Therapy in Medically Refractory Pediatric Epilepsy - Phase 1: Dosing and Tolerability Study of a Cannabidiol-Rich Whole Plant Extract of Cannabis.
Brief Title: Cannabinoid Therapy for Pediatric Epilepsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Tilray (Industry)
Responsible Party: Principal Investigator, Carter Snead, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000047417
Record Dates: First submitted 2016-11-17; First posted 2016-12-06 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): all participants will be in this arm and will receive study drug 'Cannabidiol-Rich whole Plant Extract (TIL-TC150) to assess dosing and tolerability according to study protocol.TIL-TC150 Oil is the study product The active ingredients in TIL-TC150 Oil are THC and CBD, present in a 1:50 ratio. These active ingredients are derived from Cannabis sativa L. strains produced by Tilray, and suspended in a grape seed oil. This suspension is administered at a dose of 2mg/kg/day CBD divided BID and titrated up to a maximal dose of 16mg/kg/day CBD (or maximal tolerated).
  Interventions: Drug: TIL-TC150

INTERVENTIONS:
Drug: TIL-TC150 — The active ingredients in TIL-TC150 are tetrahydrocannabinol (THC) and Cannabidiol (CBD), isolated from the Cannabis sativa L. strains produced by Tilray, and formulated into an oral liquid drug product.

SUMMARY:
This is a Phase 1 trial to determine the tolerability and optimal dose of CBD rich cannabis extract as an adjunct treatment in children with severe drug resistant epilepsy due to Dravet Syndrome. This is an open label intervention. Study duration is 20 weeks to primary analysis with continued follow-up until 64 weeks completed.

ELIGIBILITY:
Inclusion Criteria:

* Drug resistant epilepsy due to Dravet syndrome
* Must have clinically apparent seizures
* Must be able to tolerate administration of medication orally or enterally via gastrostomy tube
* Was never on Cannabinoid therapy or have not been treated with Cannabinoid products for at least last 60 days (confirmed by negative urine test for Tetrahydrocannabidiol (THC), only for those who had been treated with CBD).

Exclusion Criteria:

* Co-morbid liver or renal disease
* Without clinically-apparent seizures
* Currently taking any Cannabinoid products.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Establishment of tolerability of TIL-TC150 by measuring the number of participants with adverse events and / or abnormal laboratory values that are related to treatment | 20-64 weeks
  During this study, the dose of TIL-TC150 will be titrated according to study protocol and participant tolerance. Tolerance will be assessed as documented in title, by evaluating for adverse events clinically and by parent report of adverse event every week during the first 20 weeks of the study, also by blood work at weeks 0, 4, and between 8-16 weeks.
  For those choose to continue the study drug after 20 week period of assessment, tolerance will be evaluated by assessing for adverse events at weeks 28, 40,52 and 64.
Establishment of tolerability of TIL-TC150 by standardised side effects questionnaire -pediatric epilepsy side effects questionnaire (PESQ) | 16-64 weeks
  During this study, tolerance will also be assessed by the standardised side effects questionnaire- PESQ in clinic at weeks 2,4,8,12 and 16. For those choosing to continue therapy will be reassessed by PESQ in clinic at week 28,40,52 and 64.

SECONDARY OUTCOMES:
The impact of therapy on quality of life using the Quality of Life in Childhood Epilepsy (QOLCE) questionnaire | 16-52 weeks
  The QOLCE will be completed by parents at clinic at first visit or baseline(week 0), at maximal dose (8 weeks) and at 16 weeks for primary analysis. For those choosing to continue therapy will be reassessed at 28 weeks and 52 weeks. Parents will be provided with a research report detailing the assessment findings at study completion.
The impact of therapy on everyday behaviours using the Vineland Adaptive Behavior Scales, Second Edition. | 20-64 weeks
  Vineland Adaptive Behaviour Scale, Second Edition: is a standardized parent interview to complete either in person at the clinic or by telephone on week 0, prior to starting the TIL-TC150. The interview will also be completed again at the primary evaluation period anytime between weeks 16 and 20 and again for those choosing to continue the therapy will be reassessed during the longitudinal follow-up anytime between 52 and 64 weeks. This will be done by study team. Parents will be provided with a research report detailing the assessment findings at study completion.
change in seizure frequency from baseline | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Blathnaid McCoy, MB BCh BAO, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT02983695/Prot_SAP_000.pdf